CLINICAL TRIAL: NCT04923139
Title: Descriptive Analysis of VTE Treatment With Rivaroxaban in Japanese Clinical Practice Using a Claims Database
Brief Title: A Study to Learn About Venous Thromboembolism (VTE) Treatment With Rivaroxaban in Japanese Patients Using a Claims Database
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21471
Record Dates: First submitted 2021-06-04; First posted 2021-06-11 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Treatment of Venous Thromboembolism
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Japanese VTE patients including Ca-VTE patients: Include a large number of adult VTE patients (including Ca-VTE patients) prescribed rivaroxaban who visited facilities covered by the MDV database
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Dosage at the discretion of the treating physician

SUMMARY:
This is an observational study in which data from the past is collected for a treatment which is already available for doctors to prescribe for venous thromboembolism (VTE). VTE is a condition in which blood clots form in veins, which can lead to disability and death. This study looks at the bleeding risk in Japanese patients who are already receiving long-term rivaroxaban treatment for their VTE.

Some common causes of VTE are surgery, lack of movement, being bed-ridden and cancer. VTE that is caused by cancer is called cancer-associated venous thromboembolism (Ca-VTE).

The study treatment, rivaroxaban, is a blood thinner prescribed by doctors to help treat conditions like VTE. By thinning the blood, rivaroxaban can help keep blood flowing normally and prevent blood clots. But, rivaroxaban can lead to increased bleeding in some people.

There have been studies done in which participants with VTE and Ca-VTE received treatment with rivaroxaban for a long period of time. The overall results of those studies showed that long-term treatment with rivaroxaban helped prevent blood clots in those participants. Some of the participants had increased bleeding after this long-term treatment, while some did not. Participants with certain types of cancers, such as Ca-VTE, also had an increased risk of bleeding.

These studies, however, did not include Japanese participants. So, the researchers in this study want to learn more about the risk of bleeding in Japanese patients with VTE or Ca-VTE who receive long-term treatment with rivaroxaban. To do this, the researchers plan to use a medical database to find information for patients with VTE and Ca-VTE who have already been taking rivaroxaban for their condition. This database will help the researchers collect information about the bleeding risk of long-term rivaroxaban treatment in Japanese patients.

In this study, the researchers will learn more about:

* the characteristics of patients with VTE who are treated with rivaroxaban for a period of less than 3 months to more than 1 year
* the bleeding risk for all of the patients throughout the study
* the bleeding risk for the patients with Ca-VTE throughout the study
* the cause of any bleeding that happens

The researchers will follow and record these results for Japanese patients from October 2015 to December 2020.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of VTE recorded during the selection period (01-Apr-2016 to 31-May-2020 inclusive),
* Having a rivaroxaban prescription claim within 30 days after the VTE diagnosis ,
* Being age 18 years or older at the index date,
* Having at least 180 days baseline period.

Exclusion Criteria:

* Having evidence of atrial fibrillation, atrial flutter, dialysis, CTEPH (Chronic Thromboembolic Pulmonary Hypertension) or pregnancy during the baseline period,
* Having a claim of rivaroxaban during the baseline period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients from the Medical Data Vision Co., Ltd (MDV) extracted sample that satisfy all of the inclusion and none of the exclusion criteria will be included
Sampling Method: Non-Probability Sample
Enrollment: 2627 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Descriptive summary of bleeding risk profile of rivaroxaban, e.g.: incidence rate of / time to bleeding | Retrospective analysis from index date (first VTE diagnosis having a rivaroxaban prescription claim within 30-days after the diagnosis) up to 31-Dec-2020
  A bleeding defined as a composite of intracranial hemorrhage, intraocular bleeding, upper/lower gastrointestinal bleeding, and bleeding requiring for blood transfusion.

SECONDARY OUTCOMES:
Descriptive summary of individual components of the composite primary outcome. e.g.: incidence rate of / time to each individual components of the composite primary outcome | Retrospective analysis from index date (first VTE diagnosis having a rivaroxaban prescription claim within 30-days after the diagnosis) up to 31-Dec-2020
  Components of the composite primary outcome: intracranial hemorrhage, intraocular bleeding, upper/lower gastrointestinal bleeding, and bleeding requiring for blood transfusion.
Descriptive summary of recurrent PE/DVT event. e.g.: incidence rate of / time to recurrent PE/DVT | Retrospective analysis from index date (first VTE diagnosis having a rivaroxaban prescription claim within 30-days after the diagnosis) up to 31-Dec-2020
  PE: Pulmonary Embolism DVT: Deep Vein Thrombosis
Descriptive summary of VTE patient characteristics that treated with Rivaroxaban | Retrospective analysis from baseline period [180 days before index date (first VTE diagnosis having a rivaroxaban prescription claim within 30-days after the diagnosis)] up to 31-Dec-2020
  Patient demographic and clinical characteristics including age, gender, comorbidities, medical history and medication

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Japan databases, Japan Databases
  - Many Locations, Multiple Locations

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.